CLINICAL TRIAL: NCT07392645
Title: Clinical Efficacy of Electroacupuncture for Generalized Anxiety Disorder and Its Central Mechanism Based on Neuroimaging Changes
Brief Title: Electroacupuncture for Generalized Anxiety Disorder: Clinical Efficacy and Neuroimaging Mechanisms
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lishu Gao (Other)
Responsible Party: Sponsor-Investigator, Lishu Gao, Associate Chief Physician, First People's Hospital of Hangzhou
Organization: First People's Hospital of Hangzhou (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025KY391-1
Record Dates: First submitted 2026-01-29; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Generalized Anxiety Disorder
Keywords: Electroacupuncture; Generalized Anxiety Disorder; fMRI; Clinical Efficacy
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Electroacupuncture (EA) Group (Experimental): Paroxetine Hydrochloride Tablets + Electroacupuncture
  Interventions: Procedure: Electroacupuncture (EA); Drug: Routine Medication
- Sham Electroacupuncture (SEA) Group (Sham Comparator): Paroxetine Hydrochloride Tablets + Sham Electroacupuncture
  Interventions: Procedure: Sham Electroacupuncture (SEA); Drug: Routine Medication
- Waiting-list (WL) Group (Active Comparator): Paroxetine Hydrochloride Tablets + Delayed EA Treatment
  Interventions: Drug: Routine Medication

INTERVENTIONS:
Procedure: Electroacupuncture (EA) — Electroacupuncture (EA) is performed at acupoints including GV20 (Baihui), EX-HN1 (Sishencong), GV29 (Shenting), EX-HN16 (Anmian, bilateral), HT7 (Shenmen, bilateral), PC6 (Neiguan, bilateral), CV6 (Qihai), CV4 (Guanyuan), ST36 (Zusanli, bilateral), SP6 (Sanyinjiao, bilateral), and LR3 (Taichong, bilateral). Sterile disposable needles (φ0.18×25mm or φ0.25×40mm) are used. Electric stimulation (continuous wave, 100Hz) is applied to specific point pairs (e.g., left Sishencong + anterior Sishencong) for 30 minutes. The current intensity is adjusted to the patient's maximum tolerance. Treatment is administered 3 times per week for 4 weeks (12 sessions total).
  Arms: Electroacupuncture (EA) Group
Procedure: Sham Electroacupuncture (SEA) — Sham electroacupuncture (SEA) is performed by inserting needles into non-acupoints located 5-10 mm away from the real points used in the EA group. Shallow needling (depth of 1-2 mm) is applied. A sham EA device with a disconnected electrode lead is used; although the screen displays parameters identical to the EA group, there is no actual current output. The duration, frequency, and total number of sessions are identical to the EA group (3 times/week for 4 weeks).
  Arms: Sham Electroacupuncture (SEA) Group
Drug: Routine Medication — All groups receive Paroxetine Hydrochloride Tablets (20 mg/tablet). The initial dose is 20 mg once daily, taken orally. The daily dose may be increased in increments of 10 mg based on the patient's condition, with a minimum interval of 1 week between adjustments. The maximum daily dose is 50 mg.

SUMMARY:
This study aims to evaluate the clinical efficacy and safety of electroacupuncture (EA) in treating Generalized Anxiety Disorder (GAD). Participants will be randomly assigned to an EA group, a sham EA group, or a waiting-list control group. All participants will continue their routine medication (Paroxetine). The primary goal is to observe the reduction in anxiety symptoms using the Hamilton Anxiety Scale (HAMA). Additionally, the study will use functional MRI (fMRI) and Magnetic Resonance Spectroscopy (MRS) to explore the brain mechanisms through which EA helps alleviate anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Meet the DSM-5 diagnostic criteria for Generalized Anxiety Disorder (GAD).
* No antidepressant or anti-anxiety medication in the past 2 weeks.
* HAMA score ≥ 14.
* Right-handed（for MRI).
* Aged 18-60 years, with at least primary school education.
* Signed informed consent.

Exclusion Criteria:

* Complicated with severe cardiovascular, cerebrovascular, or organic diseases.
* History of other psychiatric disorders (e.g., schizophrenia, bipolar disorder).
* Contraindications for MRI (e.g., metal implants, claustrophobia).
* Pregnancy or lactation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 123 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Effective rate of HAMA score reduction at Week 4 | Week 4 (at the end of treatment)
  The percentage of participants who achieved a HAMA score reduction rate of ≥50% from baseline. HAMA scores are evaluated to categorize outcomes as recovered, markedly effective, effective, or ineffective.

SECONDARY OUTCOMES:
Change from Baseline in Hamilton Anxiety Scale (HAMA) Scores | Baseline, Week 2, Week 4, and Week 8
  HAMA is used to assess the severity of anxiety symptoms. It contains 14 items, including somatic and psychic anxiety. Total scores range from 0 to 56, where higher scores indicate more severe anxiety
Change from Baseline in Social Disability Screening Schedule (SDSS) Scores | Baseline, Week 2, Week 4, and Week 8
  SDSS is used to evaluate the daily functioning of patients. It consists of 10 items, with each item scored from 0 to 2. Higher total scores reflect a higher degree of social disability.
Frequency of Participants with Changes in Paroxetine Dosage | Week 2, Week 4, and Week 8
  The study will record whether the daily dose of Paroxetine increased, remained unchanged, or decreased compared to the baseline.
Treatment Emergent Symptom Scale (TESS) Scores | Week 2, Week 4, and Week 8
  TESS is used to evaluate adverse reactions to psychiatric medications, covering symptom severity, relationship with the drug, and measures taken.
Changes in Functional Connectivity (FC), Regional Homogeneity (ReHo), and Amplitude of Low-Frequency Fluctuation (ALFF) | Baseline and Week 4
  Twenty right-handed subjects will be randomly sampled from each group for the neuroimaging mechanism study. Resting-state functional MRI (fMRI) will be used to analyze brain activity changes. FC describes the synchronization between different brain regions; ReHo and ALFF describe the local homogeneity and intensity of brain activity. Resting-state functional MRI (fMRI) will be used to analyze brain activity changes. FC describes the synchronization between different brain regions; ReHo and ALFF describe the local homogeneity and intensity of brain activity.
Changes in Brain Metabolite Concentrations via Magnetic Resonance Spectroscopy (MRS) | Baseline and Week 4
  Twenty right-handed subjects will be randomly sampled from each group for the neuroimaging mechanism study. 3D 1H-MRS will be used to measure the absolute concentrations of neurotransmitters in ROI (amygdala, hypothalamus, etc.), e.g. 5-HT, NE, DA, GABA, and CRF

IPD SHARING:
Plan to Share IPD: No